CLINICAL TRIAL: NCT06176417
Title: Horizontal Ridge Augmentation Using Decompression Technique Versus Ridge Splitting in Atrophic Posterior Mandibular Ridge With Simultaneous Implant Placement
Brief Title: Comparison Between Different Horizontal Ridge Augmentation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sara elmaghraby, assistant lecturer of oral and maxillofacial surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A03030821
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Atrophic Ridge

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Eight implants were placed in patients of missing single tooth / teeth in posterior mandible with subsequent horizontal ridge augmentation by decompression technique.
  Interventions: Procedure: horizontal ridge augmentation by decompression technique.
- group 2 (Experimental): Eight implants were placed in patients of missing single tooth / teeth in posterior mandible with subsequent horizontal ridge augmentation by ridge splitting technique using piezosurgery.
  Interventions: Procedure: horizontal ridge augmentation by ridge splitting technique using piezosurgery.

INTERVENTIONS:
Procedure: horizontal ridge augmentation by decompression technique. — Instead of a cover screw, a 2-mm healing abutment was used after implant insertion
  Arms: group 1
Procedure: horizontal ridge augmentation by ridge splitting technique using piezosurgery. — horizontal ridge augmentation was done using piezosurgery tips and bone expanders
  Arms: group 2

SUMMARY:
Sixteen patients were selected from the Outpatient Clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University for replacement of missed single tooth / teeth in posterior atrophic mandible by dental implant.

Patients' grouping:

Patients were divided randomly into two equal uniform groups as follow:

Group I:

Eight implants were placed in patients of missing single tooth / teeth in posterior mandible with subsequent horizontal ridge augmentation by decompression technique.

Group II:

Eight implants were placed in patients of missing single tooth / teeth in posterior mandible with subsequent horizontal ridge augmentation by ridge splitting technique using piezosurgery.

All patients were evaluated clinically and radiographically at regular time interval immediately, 6 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient's cooperation, motivation and good oral hygiene.
* Patient medically free from systemic diseases that absolutely contraindicate implant surgery.
* Moderately atrophic posterior mandible (horizontal alveolar dimension is not more than 4 mm at the crest), with minimum 10 mm vertical height.
* Patients prepared to comply with the follow-up and maintenance programme.
* Free from history of bruxism / parafunctional habits.

Exclusion Criteria:

* Patients with local pathological disease such as cyst, tumor at the planned surgical site.
* Pregnant patients.
* Heavy smoker patients.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-08-26 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge width | 12 months
  The ridge width was measured on the cross section view at different time interval from the outer surface of the buccal bone to the outer surface of the lingual bone perpendicular to the line marking the long axis of the implant at implant platform.
  Changes in alveolar ridge width was measured by subtracting ridge width value after 6 and 12 months from immediate postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Elmagraby, Al Mansurah, Egypt